CLINICAL TRIAL: NCT02932761
Title: Comparison of the Therapeutic Effects of Vaginal Repair and Vaginal Repair Combined With GnRHa in the Treatment of Cesarean Scar Diverticula: a Randomized Clinical Trial
Brief Title: Comparison of the Therapeutic Effects of VR and VR + GnRHa in the Treatment of Cesarean Scar Diverticula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xipeng Wang (Other)
Responsible Party: Sponsor-Investigator, Xipeng Wang, Professor, Shanghai First Maternity and Infant Hospital
Organization: Shanghai First Maternity and Infant Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSD-001
Record Dates: First submitted 2016-10-08; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Cesarean Scar Diverticula
Keywords: cesarean scar diverticula; vaginal repair; GnRHa
MeSH Terms: interventions — Goserelin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VR + GnRHa (Experimental): CSD patients were treated with vaginal repair of CSD in combination with GnRHa (Zoladex, 3.6 mg, AstraZeneca, Macclesfield, United Kingdom) as a subcutaneous injection (abbreviated as VR + GnRHa). In the group of VR + GnRHa, 2 doses of GnRHa were administered. The first dose was injected at the time of hysteroscopy examination, and the second dose was administered one day after the VR surgical procedure. The detailed procedure of VR has been described in our previous study (Zhou et al., 2016).
  Interventions: Drug: GnRHa; Procedure: Vaginal repair of CSD
- VR (Placebo Comparator): CSD patients were treated with vaginal repair of CSD in combination with 0.01 ml saline as a subcutaneous injection (abbreviated as VR). In the group of VR, 2 doses of saline were administered. The first dose was injected at the time of hysteroscopy examination, and the second dose was administered one day after the VR surgical procedure. The detailed procedure of VR has been described in our previous study (Zhou et al., 2016).
  Interventions: Procedure: Vaginal repair of CSD

INTERVENTIONS:
Drug: GnRHa — Two doses of GnRHa were administered by subcutaneous injection. The first dose was injected at the time of hysteroscopy examination, and the second dose was administered one day after the VR surgical procedure.
  Other Names: Zoladex, 3.6 mg, AstraZeneca, Macclesfield, United Kingdom
  Arms: VR + GnRHa
Procedure: Vaginal repair of CSD — The procedure of vaginal repair of CSD was shown as following. The bladder was dissected away carefully from the uterus toward the abdominal cavity until the peritoneum was reached. The CSD tissue was cut to the normal healthy muscle after the abdominal cavity had been entered, and the lower uterine segments had been completely exposed. A double layer of 1-0 absorbable interrupted sutures was used to close the incisions.

SUMMARY:
Cesarean scar diverticula (CSD) is a novel recognized cause of postmenstrual abnormal uterine bleeding in women. No clinical guidelines have been issued for the management of CSD. The investigators have previously demonstrated that vaginal repair of CSD was an relative effective treatment of CSD. However, only 28.2% of the CSD patients normalized to less than 7 days of menstruation, whereas 51.2% of women had 7 to 10 days of menstruation at 6 months post vaginal repair. Postoperative menstruation may contribute to surgical site infections, which may subsequently affect the healing of uterine scars. Treatment CSD patients with gonadotropin-releasing hormone agonist (GnRHa) may has the potential to improve therapeutic effects of vaginal repair. Therefore, the current multiple-center randomized controlled trial was designed to evaluate whether the application of GnRHa in combination with vaginal repair could achieve better clinical effects than those achieved by vaginal CSD repair alone.

DETAILED DESCRIPTION:
Postoperative menstruation may contribute to surgical site infections, an inflammatory environment, congestion at the site of the suture, immune cell infiltration, and other effects and may subsequently affect the healing of uterine scars. It is reasonable to hypothesize that delaying the postoperative menstrual recovery period may allow uterine scars to heal without the inflammatory reaction caused by menstruation. Treatment with gonadotropin-releasing hormone agonist (GnRHa) has the ability to suppress follicle-stimulating hormone (FSH) and luteinizing hormone (LH) release, thereby maintaining low estrogen levels and causing temporary amenorrhea. A prolonged menstrual recovery period may be achieved after GnRHa administration. Vaginal repair of CSD combined with GnRHa may improve the therapeutic effects of treatment of CSD. Therefore, the randomized study was designed to evaluate whether the application of GnRHa in combination with vaginal repair could achieve better clinical effects than those achieved by vaginal CSD repair alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are younger than 40.
2. Clearly diagnosed with CSD.
3. Experiencing clinical features of abnormal uterine bleeding, prolonged menstrual flow (the duration of menstruation is more than 7 days).
4. The thickness of the remaining muscular layer of CSD was less than 3 mm.
5. The women are at least 20 years old with singleton pregnancies and had undergone a cesarean delivery after at least 37 weeks of gestation.
6. The medicine conservative treatment is invalid.
7. Refusing or use birth control pills contraindications.
8. No serious medical problems (important viscera function in the normal range).
9. No uterine fibroids, endometriosis, adenomyosis, and patients with ovarian cysts.
10. No gynaecology or other malignant tumors.
11. Sign the informed consent.

Exclusion Criteria:

1. Over the age of 40;
2. Indefinite diagnosis.
3. The absence of clinical manifestations of CSD.
4. The presence of menstrual irregularities before cesarean delivery.
5. Coagulation disorders.
6. Malignant tumors.
7. With severe medical problems (severe liver disease, kidney disease, respiratory diseases, heart disease or uncontrolled diabetes, epilepsy, etc., dysfunction of important organs).
8. Known chronic inflammatory diseases, any other uterine diseases (such as uterine fibroids, endometriosis and adenomyosis), uterine surgery except cesarean section.
9. Use of intrauterine devices.
10. Unwilling to comply with the research plan.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
thickness of the remaining muscular layer (mm) | 6 months after vaginal repair of CSD
  The thickness of the remaining muscular layer is measured by transvaginal ultrasound.
duration of menstruation (day) | 6 months after vaginal repair of CSD
  The menstruation duration in CSD patients is collected 6 months after vaginal repair of CSD.

SECONDARY OUTCOMES:
the length of CSD (mm) | 6 months after vaginal repair of CSD
  The length of CSD is measured by transvaginal ultrasound.
the width of CSD (mm) | 6 months after vaginal repair of CSD
  The width of CSD is measured by transvaginal ultrasound.
the depth of CSD (mm) | 6 months after vaginal repair of CSD
  The depth of CSD is measured by transvaginal ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Xipeng Wang, M.D., Ph.D.,, Study Chair — Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University
Locations (1):
- Department of Gynecology, Shanghai First Maternity and Infant Hospital, affiliated to Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No